CLINICAL TRIAL: NCT05590026
Title: Pediatric Pectointercostal and ESP Block in Cardiac Surgery Surgery
Brief Title: Pediatric Pectointercostal and ESP Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, ebru biricik, Associate Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pediatric Pectointercostal
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pectointercostal and ESP block (Active Comparator): Pectointercostal and ESP block will apply to the children after intubation. Totally bupivacain %0.25, 2.5 mg/kg will apply.
  Interventions: Drug: Pectointercostal and ESP block
- No Block (Placebo Comparator): No block will apply to the patient
  Interventions: Drug: Pectointercostal and ESP block

INTERVENTIONS:
Drug: Pectointercostal and ESP block — Both Pectointercostal at between 4th and 5th costa and ESP block will apply at thoracal 6 level to the patient.
  Other Names: Fascia plane blocks

SUMMARY:
American Society of Anaesthesiologist physical status II-III, aged between 2, 12 patients which underwent open cardiac surgery will recruited to this study. These subjects will Ultrasound (USG) guided erector spinae block will perform at T6 level (bilaterally) and pectointercostal plane block at 4-5 intercostal space to the all patient under general anaesthesia. Totally bupivacaine %0.25 2.5 mg/kg will use blocks. 2 ml %0.25 bupivacain will apply to the chest tube area at the end of surgery. 0.1 microgram/kg morphine will apply intravenously at last 30 minutes of surgery postoperative analgesia to all patients. Postoperative pain and agitation assessment will perform with FLACC and Watcha scores

DETAILED DESCRIPTION:
American Society of Anaesthesiologist physical status II-III, aged between 2-12, 60 patients which underwent open cardiac surgery will recruited to this study. The patients were randomly allocated into two groups (1:1), via a computer-generated randomization list. Ultrasound (USG) guided erector spinae block will perform at T6 level (bilaterally) and pectointercostal plane block at 4-5 intercostal space to the 30 patients under general anaesthesia in Group block and block will not perform to the control group. Sevoflurane+remifentanil and O2/air combination will perform to the all patients during the surgery. Totally bupivacaine %0.25 2.5 mg/kg will use for blocks.2 ml %0.25 bupivacain will apply to the chest tube area at the end of surgery. 0.1 microgram/kg morphine intravenously will apply for postoperative analgesia to the all patients at last 30 minutes of surgery. Postoperative pain and agitation assessment will perform with FLACC and Watcha scores. FLACC, Watcha scores, morphine consumption and complications will record.Paracetamol 10 mg/kg will repeat to the all patients at the 12th of postoperative period, intravenously. The patient controlled anesthesia with morphin will apply to the all patients. If the FLACC score is higher than 4, morphine 0.015 mg/kg will administer intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 2-12 years
* ASA II-III children
* The children who undergoing open heart surgery

Exclusion Criteria:

* Coagulopaty
* Allergy of local anesthetic
* Liver and renal failure
* Obesity (BMI >35kg/m2)
* Infection at the block area

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative analgesia | 24 hours in Postanesthesia care unit (PACU)
  Postoperative analgesia will asses Face, Legs, Activity, Cry, Consolability (FLACC) score in (Postanesthesia care unit) PACU till the 24th hours postoperatively. FLACC score reflects pain score between 0-10. 0 means zero pain, 10 means worse pain score
Postoperative morphine consumption | 24 hours in Postanesthesia care unit (PACU)
  Postoperative morphine consumption will record till the postoperative 24 th hours

SECONDARY OUTCOMES:
Postoperative agitation | First 24 hours at Postanesthesia care unit (PACU)
  The patients will asses with Watcha score for postoperative agitation in Postanesthesia care unit (PACU) till the postoperative 24th hours. Watcha score reflects delirium score (scale between 0 to 4). A child with a score of >2 on the Watcha score can be considered to have emergence delirium. (Points between 0-4) Watcah is one of the author's name.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Biricik, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No